CLINICAL TRIAL: NCT01487590
Title: A Simple Blind Controlled Randomized Trial: Cephalic Version by Acupuncture-moxibustion vs Placebo for Breech Presentation
Brief Title: Cephalic Version by Acupuncture-Moxibustion for Breech Presentation
Acronym: ACUVERSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DGS 2006/0404
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breech Presentation
Keywords: pregnancy; breech; acupuncture; moxibustion; version
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture moxibustion (Active Comparator): Six interventions with acupuncture moxibustion, stimulating point BL67, during 20 minutes each, 48 hours apart.
  Interventions: Other: Acupuncture moxibustion
- Placebo (Placebo Comparator): Six interventions with placebo (inactivated laser), stimulating point BL67, during 20 minutes each, 48 hours apart
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Acupuncture moxibustion — Six interventions with acupuncture moxibustion, stimulating point BL67, during 20 minutes each, 48 hours apart.
  Other Names: no applicable
  Arms: Acupuncture moxibustion
Other: Placebo — Six interventions with placebo (inactivated laser), stimulating point BL67, during 20 minutes each, 48 hours apart
  Other Names: no applicable
  Arms: Placebo

SUMMARY:
For breech presentation, the cesarean section rate is decreased by external cephalic version. This is a painful operation, with some rare but serious complications. The aim of this trial is to evaluate the effectiveness of acupuncture-moxibustion, a non-invasive technique, to correct breech presentation before 37 weeks of gestation.

DETAILED DESCRIPTION:
Monocentric controlled randomized trial in a simple blind fashion, comparing acupuncture-moxibustion versus a placebo in singleton pregnancies with breech presentation between 33+5 to 35+5 weeks of gestation. The intervention arm consists of acupuncture-moxibustion at the BL67 acupuncture point, for six seances of twenty minutes two days apart. In the placebo group, the cold light of an inactivated laser is to be applied in the same point during the same time. When cephalic version fail, a manual external cephalic version is to be proposed. The main outcome measure is cephalic presentation at 37+2 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* breech presentation,
* SINGLETON

Exclusion Criteria:

* maternal age between 18 ans 45,
* multiple gestation,
* fetal or uterine malformation,
* premature rupture of membranes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cephalic presentation | at 37+2 weeks of gestation
  Each participant women will be examined at 37+2 weeks to determine the fetal presentation. Ultrasonography will be performed in case of doubt.

SECONDARY OUTCOMES:
Successful manual external cephalic version after intervention | Before 41 weeks of gestation
  In case of failure of acupuncture/moxibustion or placebo, the success of manual external cephalic version will be studied.
Cephalic presentation at delivery | Date of delivery
  The rate of cephalic presentation at delivery will be described
Cesarean section rate | Date of delivery
  The cesarean section rate will be described
Premature rupture of membranes | Before delivery
  The rate of premature rupture of membranes will be described

CONTACTS AND LOCATIONS:
Overall Officials: Damien SUBTIL, PhD-MD, Principal Investigator — CHRU de Lille, France; Capucine COULON, MD, Study Chair — CHRU de Lille, France
Locations (1):
- Hopital Jeanne de Flandre, CHRU de Lille, Lille, France

REFERENCES:
- [Result] Coulon C, Poleszczuk M, Paty-Montaigne MH, Gascard C, Gay C, Houfflin-Debarge V, Subtil D. Version of breech fetuses by moxibustion with acupuncture: a randomized controlled trial. Obstet Gynecol. 2014 Jul;124(1):32-39. doi: 10.1097/AOG.0000000000000303. PMID 24901279